CLINICAL TRIAL: NCT01610908
Title: A Multicenter Randomized Controlled Trial to Compare the Effect of Schroth Exercises to Standard Care on Curve Characteristics, Posture, and Quality Of Life in Adolescents With Idiopathic Scoliosis
Brief Title: Multicenter Schroth Exercise Trial for Scoliosis
Acronym: MultiSETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Glenrose Foundation (Other); Scoliosis Research Society (Other); SickKids Foundation CIHR Institute of Human Development, Child and Youth Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00043397
Record Dates: First submitted 2012-04-02; First posted 2012-06-04 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Scoliosis
Keywords: Adolescent; Idiopathic; Scoliosis; Schroth; Exercises; Conservative treatment
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Schroth exercises (Experimental): The experimental group receives the Schroth exercises treatment.Patients in this arm receive 5 individual sessions with a Schroth therapist for introduction to the approach. They they receive a home program consisting of 3-4 exercises to do at home everyday for 30-45 minutes. They come to weekly group therapy sessions to where exercise prescription is adjusted.
  Interventions: Other: The Schroth exercises treatment
- Standard of care (No Intervention): "The Standard of care" is a control group that will continue receiving the standard North American treatment prescribed by a surgeon (observation or brace [if meeting SRS criteria]) for of 6 months. After 6 months, the participants will receive the Schroth exercises intervention for 6 months.
- Global Postural Re-education (Montréal) (Active Comparator): The active group (in Montréal only) receives the Global Postural Re-Education exercises treatment.Patients in this arm come to weekly individual 1 hour long therapy sessions where exercise prescription is adjusted. Selection of posture exercises is based on scoliosis type, on muscular chain stiffness associated with posture alterations and on position increasing scoliosis or pain (lying, sitting, standing).
  They they receive a 15-min home program consisting of 1 to 2 exercises to do at home everyday.
  Interventions: Other: Global Postural Re-Education

INTERVENTIONS:
Other: The Schroth exercises treatment — The Schroth approach consists of 3D scoliosis-specific exercises based on sensorimotor and kinesthetic principles. The goal of Schroth exercises is to teach patients to consciously maintain the correct posture in daily living activities in order to improve the curve, pain, and self-image. To achieve this goal, Schroth exercises focus on endurance and strength training of postural muscles. Schroth exercises also aim to improve posture motor control by repeating corrective movements with progressively less feedback and less passive support.
  Dosage: 5 individual 1-hour long sessions, continued with the daily 45 minutes home exercise program. In addition, patients are required to come weekly for 1-hour long group sessions over the span of 6 months.
  Other Names: Scoliosis specific exercises.; The Schroth Approach.
  Arms: Schroth exercises
Other: Global Postural Re-Education — The 6-month supervised Global Postural Re-education intervention involves active movements and postures aimed at realigning joints, stretching shortened muscles and enhancing the contraction of antagonist muscles, thus avoiding postural asymmetry. These postures imply an active participation of the patient. Global Postural Re-education includes eight therapeutic postures, lying, sitting or standing, held for 15/20 min. each. Variously combinations are used during sessions chosen on based on the amount of pain, load capacity, age of the patient, and muscle chains to be stretched. Static and dynamic functions are also employed for about five minutes each sessions to use the recovered flexibility in functional activities Dosage: Weekly individual 1-hour long sessions, with daily 15 minutes home exercise program over 6 months.
  Other Names: GPR; Ré-éducation posturale globale
  Arms: Global Postural Re-education (Montréal)

SUMMARY:
The primary aim of this multicenter randomized controlled trial is to compare the effect of a 6 month "Schroth exercise program combined with standard-of-care" to "standard-of-care alone" on scoliosis curve severity measured using the Cobb angle.

Secondary aims include:

1. To determine the effect of Schroth exercises at 6 months on secondary outcomes including quality-of-life, spinal appearance, objective posture and spinal muscle endurance measurements.
2. To determine the efficacy of 6 months of Schroth therapy offered to control participants after completing 6 months in the standard-of care group (using subjects as their own controls)
3. To determine if the effects of the 6 months supervised Schroth exercise program can be maintained after supervised therapy is terminated.

At Hopital Ste-Justine, the following secondary aims will be pursued to examine the preliminary evidence about the effect of Global Postural Re-education (to satisfy the local ethics committee request because Global Postural Re-education exercises were offered routinely to patients at that institution prior to the trial).

A. To compare the effect and to quantify the treatment effect sizes of 6 months of "Global Postural Re-education exercises with North American standard Care consisting of only observation and bracing" to "Schroth exercises combined with North American standard care" and to "North American standard care alone" on scoliosis curve severity measured using the Cobb angle.

B. To estimate the effect and quantify the treatment effect sizes of 6 months of "Global Postural Re-education exercises with North American standard Care" to "Schroth exercises combined with North American standard care" and to "North American standard care alone" on outcomes including quality-of-life, perceived spinal appearance, objective posture and spinal muscle endurance measurements.

C. To determine if the effects of "Global Postural Re-education exercises with North American standard Care" can be maintained after discontinuing supervision.

D. To estimate the feasibility of conducting a randomized trial focused on Global Postural Re-education exercises by quantifying enrollment rates, attendance at scheduled exercise sessions and compliance with the home exercises prescribed.

DETAILED DESCRIPTION:
Multicenter Schroth Exercise Trial for Scoliosis (SETS study) Adolescent Idiopathic Scoliosis (AIS) is a progressive 3D deformity of the spine. It is the most common orthopedic condition in adolescents. Of those with curves larger than 10°, 90% are females. Scoliosis often results in chronic pain, poor posture, function, and self-image.

Curves greater than 30° are braced or later surgically corrected. In Europe but not the Americas, small curves (<30°) are treated with exercises to prevent the need for bracing and moderate curves with bracing and exercises to prevent surgery. Bracing is uncomfortable and patients fear surgery. In contrast, exercises are generally well received.

Schroth exercises are the most studied scoliosis exercises and have achieved very good outcomes. Schroth was the first exercise approach to offer formal certification training. No randomized controlled trial has focused on the Schroth method. Only 1 randomized controlled trial and only 3 prospective controlled studies with important methodological flaws were included in a recent review of the effect of all types of scoliosis exercises that found that exercises slowed the worsening of scoliosis. A randomized controlled trial on Schroth exercises is needed.

Schroth exercises are asymmetric scoliosis-specific postural exercises and aim to improve the curve, posture, pain, function, and self-image. Schroth exercises target endurance and strength training of the abdominal, back, and leg muscles. Schroth exercises also aim to improve motor control of the posture by repeating corrective movements with progressively less feedback.

Objectives: (1) To compare the effect of 6 month "of Schroth exercises combined with standard-of-care" to "standard-of-care alone" on scoliosis curve severity measured using the Cobb angle.

Secondary aims include determining treatment effects on quality-of-life, spinal appearance, posture and spinal muscle endurance and monitoring if effect are maintained at long-term follow-ups.

See above for objectives corresponding to the secondary analysis planned at Hopital Ste-Justine.

Methodology:

Participants: Two hundred fifty-eight females with AIS will be recruited for this study from our scoliosis clinic. Females 10-16 years old with curves 10° to 45°, and Risser less than or equal to 3 will be included. Patients who are planning surgery, have had surgery, worn a brace or to be discharged will be excluded.

Procedures: Participants will be randomized to the standard-of-care group (observation of bracing if Boston brace criteria are met) or the Schroth exercise treatment group.

(At hospital Ste-Justine, only because of the ethics committee requested we include a third trial arm, we will randomize an equal number of subjects to each of the three trial arms (Global Postural Re-education, Schroth and Standard care) using the a variable blocked randomization specific to this site. This implies recruiting an estimated additional 52 patients to be randomized to the Global Postural Re-education group.) Outcomes will be measured by evaluators blind to randomization status at baseline and at 3 and 6 month follow-ups. The primary outcome is the spinal curvature angle on radiograph at 6 months. Secondary outcomes analyzed at 3, and 6 months include radiographs (Cobb angle, rotation), Scoliosis Research Society-22r quality-of-life domain scores (self-image, function, pain), spinal appearance questionnaire domain scores, postural measures (surface topography), and Sørensen back muscle endurance. Radiographs and Scoliosis Research Society-22 measures from routine scoliosis clinic visits will also be obtained from the clinic database until discharged from routine care. Measurement properties of all measures are adequate.

Standard-of-care subjects will be under observation or treated with bracing if they meet the Scoliosis Research Society bracing criteria for 6 months and then be offered the Schroth exercise treatment as a recruitment incentive necessary based on our pilot. Treated patients will receive supervised and standardized Schroth exercises combined with a home program in addition to standard of care for 6 months. Parents will be involved to enhance (and monitor) compliance. (At hôpital Ste-Justine only, one group will receive the 6-month supervised Global Postural Re-education intervention consisting of individual training sessions with a therapist combined with a home exercise program consisting of 1 or 2 exercises to perform twice weekly in addition the standard of care).

Analyses: Linear mixed models will be used to assess differences in group changes from baseline, to 3 months and 6-month, and adjusting for relevant covariates (including age, and risk of progression).

Expected findings: Schroth exercises will improve curve characteristics, quality of life, posture, pain, and muscular endurance in patients with adolescent idiopathic scoliosis. The study team is integrated within the Edmonton scoliosis clinic, Montréal's Centre Hospitalier Universitaire Ste-Justine clinic and Calgary's Alberta Children Hospital Clinic. Research results can directly influence practice.

ELIGIBILITY:
Inclusion Criteria:

* adolescent idiopathic scoliosis
* Females
* 10° to 45° according to Cobb (scoliosis curve)
* with or without a brace
* ability to travel weekly to our lab
* skeletal maturity measured by Risser (0-3)

Exclusion Criteria:

* other type of scoliosis
* patients with curves > 50°
* surgical candidates
* patients who have had a corrective spinal surgery
* out-of town candidates, without possibility to travel to our lab

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2011-04; Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Cobb angle | From baseline to 6 months
  The angle from a posterior anterior full spine radiographs between the upper endplate of the upper end vertebra of the largest curve and the lower endplate of the lower end vertebra from the largest curve.

SECONDARY OUTCOMES:
Change in Vertebral rotation | Change from baseline to 6 months
  Using a posterior-anterior radiograph and a semi-automated algorithm in Matlab the rotation of the most rotated vertebra in the curve will be extracted. The algorithm relies on the semi-automated identification of the position of the the pedicles vs the edges of the vertebral body.
Change in Back muscle endurance | From baseline, to 3 months and to 6 months follow-ups
  Using Sørensen back muscle endurance test, we record the time until fatigue to maintain the torso unsupported from the waist up horizontally against gravity with the arms crossed against the chest and the head and neck maintained aligned with the trunk. Leg are maintained firmly against the bed using gait belts tightened against a treatment table. The test stops if patients lose the ability to maintain the position after one reminder for good form or if they personally ask to stop because of pain or fatigue.
Change in Scoliosis Research Society-22r questionnaire scores | From baseline, to 3 months and to 6 months follow-ups
  The Scoliosis Research Society-22r questionnaire is available from SRS.org. It is a self-reported tools assessing self-image, function, pain, mental health with 5 questions each and satisfaction with care with 2 questions. A total score is also available based on all 22 questions.
Change in Spinal Appearance Questionnaire scores | From baseline, to 3, and to 6 months
  The Spinal Appearance Questionnaire measures patients' perception of their spinal deformity using standardized drawings and questions.
  The new version of the Spinal Appearance Questionnaire containing 20 items will be used in this study, which addresses the following domains: General (items 9, 10, and 19), Curve (item 1), Prominence (items 2 and 3), Trunk shift (item 4 and 5), Waist (items 11, 12, and 13), Shoulders (items 6 and 16), Kyphosis (item 7), Chest (items 14 and 15) and Surgical scar (item 17). In scoring, we will use all domains, except Kyphosis and Surgical scar, because these domains are not relevant to the subjects in this study.
Global rating of change relative to baseline | at 3 and at 6 months
  A 15-point global rating scale will be used to assess the patient's perceived change over time. The scale ranges from -7 (a very great deal worse) to +7 (a very great deal better).
Change in Self-efficacy | From baseline, to 3 and to 6 months
  This questionnaire measures self-efficacy for overcoming barriers to physical activity (defined as corrective exercise activities) using 8 items rated from 1 (Disagree a lot) to 5 (Agree a lot).
Change in numeric pain ratings and diagram | From baseline, to 3 and to 6 months
  A scale from 0 (no pain) to 10 (worst imaginable pain) will assess current, best, worst pain intensity in the last 24 hours. A body pain diagram will help categorize the location of symptoms.
Change in surface topography assessment of posture | From baseline, to 3 and to 6 months
  Four Laser Scanners (Edmonton) and 4 optical scanners ( Montréal and Calgary) are used to capture full-torso scans. Subjects are positioned in a standard frame, and 18 reference points marked. Parameters are extracted by digitizing 15 landmarks. Parameters quantifying the external back surface deformity are: decompensation, cosmetic score (combines the shoulder angle, scapula angle and waist asymmetry), in the coronal plane, the deformity in the axial plane index, Hump Sum, trunk twist in the transverse plane and kyphotic and lumbar angles in the sagittal plane.
  From full torso scans are: lateral deviation of centroid, and back surface rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Parent, PT, MSc, PhD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Alberta Children Hospital, Calgary, Alberta
  - University of Alberta, Faculty of Rehabilitation Medicine, Dept. Physical Therapy, Edmonton, Alberta
  - CHU Ste-Justine, Montreal, Quebec

REFERENCES:
- [Background] Watkins E, Bosnjak S, Parent E. Algorithms to prescribe Schroth exercises for each of four Schroth curve types. Scoliosis. 2012 Jan 27;7 Suppl 1:P22.
- [Background] Schreiber S, Parent E, Watkins E, Hedden D. An algorithm for determining scoliosis curve type according to Schroth. Scoliosis. 2012 Jan 27;7 Suppl 1:O53.
- [Background] Schreiber S, Parent EC, Hedden DM, Moreau M, Hill D, Lou E. Effect of Schroth exercises on curve characteristics and clinical outcomes in adolescent idiopathic scoliosis: protocol for a multicentre randomised controlled trial. J Physiother. 2014 Dec;60(4):234; discussion 234. doi: 10.1016/j.jphys.2014.08.005. Epub 2014 Oct 17. PMID 25439713
- [Background] Schreiber S, Parent E, Khodayari Moez E, Hedden D, Hill D, Moreau M, Lou E, Watkins E, Southon S. (2016). Schroth Physiotherapeutic Scoliosis-specific exercises improve Cobb Angles in adolescents with Idiopathic Scoliosis - a randomized controlled trial.10th Annual WCHRI Research Day, Edmonton Canada, (oral 23 Page 27)
- [Background] Schreiber S, Parent EC, Moez EK, Hedden DM, Hill D, Moreau MJ, Lou E, Watkins EM, Southon SC. The effect of Schroth exercises added to the standard of care on the quality of life and muscle endurance in adolescents with idiopathic scoliosis-an assessor and statistician blinded randomized controlled trial: "SOSORT 2015 Award Winner". Scoliosis. 2015 Sep 18;10:24. doi: 10.1186/s13013-015-0048-5. eCollection 2015. PMID 26413145
- [Result] Parent EC, Schreiber S, Hedden D, Moreau M. The effect of a 6-month Schroth exercise program: a pilot study using subjects as their own controls. Scoliosis. 2013;8(Suppl 2):045.
- [Result] Schreiber S, Parent EC, Hedden DM, Moreau M, Hill D, Watkins EM. The effects of a 6-month Schroth intervention for Adolescent Idiopathic Scoliosis (AIS): preliminary analysis of an ongoing randomized controlled trial. Scoliosis. 2013;8(Suppl 2):O44.
- [Result] Schreiber S, Parent E, Hedden D, Moreau MJ. Clinical Significance of The Effect of A Six-Months Schroth Exercise Intervention in Adolescents with Idiopathic Scoliosis. 2015 Annual Meeting Pediatric Orthopaedic Society of North America (POSNA), e-poster #18, p391, 2015
- [Result] Schreiber S, Parent EC, Hill DL, Hedden DM, Moreau MJ, Southon SC. Schroth physiotherapeutic scoliosis-specific exercises for adolescent idiopathic scoliosis: how many patients require treatment to prevent one deterioration? - results from a randomized controlled trial - "SOSORT 2017 Award Winner". Scoliosis Spinal Disord. 2017 Nov 14;12:26. doi: 10.1186/s13013-017-0137-8. eCollection 2017. PMID 29164179
- [Result] Schreiber S, Parent EC, Khodayari Moez E, Hedden DM, Hill DL, Moreau M, Lou E, Watkins EM, Southon SC. Schroth Physiotherapeutic Scoliosis-Specific Exercises Added to the Standard of Care Lead to Better Cobb Angle Outcomes in Adolescents with Idiopathic Scoliosis - an Assessor and Statistician Blinded Randomized Controlled Trial. PLoS One. 2016 Dec 29;11(12):e0168746. doi: 10.1371/journal.pone.0168746. eCollection 2016. PMID 28033399
- [Result] Schreiber S**, Parent EC, Hill DL, Hedden DM, Moreau M, Southon S. (2018). How much change in the Cobb angle is needed for the patients to observe positive change in their backs following a Schroth intervention? In Abstract Book Program from XIII International Meeting of the Society for Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT), Dubrovnik, Croatia, April 19-21, 2018, P71. (Winner of the 2018 SOSORT Award)
- [Result] Schreiber S*, Parent E, Hill D, Hedden D, Moreau M, Southon S. (2017). Schroth Physiotherapeutic Scoliosis-Specific Exercises for Adolescent Idiopathic Scoliosis: How Many Patients Require Treatment To Prevent One Deterioration?. Book of abstracts of the 12th International Meeting of the International Society on Scoliosis Orthopaedic and Rehabilitation Treatment. Lyon, France, May 4 to 6 2017, O37.66, S7110-111
- [Result] Schreiber S*, Parent EC, Moez EK, Hedden DM, Hill D, Moreau M, Lou E, Watkins EM*, Southon SC. (2016). The effect of Schroth exercises added to the standard of care on the Cobb angle in adolescents with idiopathic scoliosis: An assessor and statistician blinded randomized controlled trial Scoliosis and Spinal Disorders 2017 12(Suppl 1):17 O60. Proceedings of The First Joint Meeting of the International Research Society of Spinal Deformities and the Society on Scoliosis Orthopaedic and Rehabilitation Treatment, Banff, Alberta, Canada, May 25-28, 2016. Paper O-81, pages 68-69
- [Result] Schreiber S*, Parent EC, Hedden DM, Hill DL Scoliosis and Spinal Disorders 2017 12(Suppl 1):17 O70. (2016). Minimal important differences in Scoliosis Research Society-22R, Spinal Appearance Questionnaire, Cobb angle and Biering-Sorensen back muscle endurance test following a six-month Schroth exercises intervention in adolescents with idiopathic scoliosis. Proceedings of The First Joint Meeting of the International Research Society of Spinal Deformities and the Society on Scoliosis Orthopaedic and Rehabilitation Treatment, Banff, Alberta, Canada, May 25-28, 2016. Paper 0-93, pages
- [Result] Parent EC, Schreiber S*, Moez EK, Preston S*, Hedden D, Moreau M, Hill D, Southon S, Watkins E*. (2016). Effects of Schroth exercises added to standard care in adolescents with idiopathic scoliosis (AIS) on surface topography parameters: A randomized controlled trial (RCT) Scoliosis and Spinal Disorders 2017 12(Suppl 1):17 O61. Proceedings of The First Joint Meeting of the International Research Society of Spinal Deformities and the Society on Scoliosis Orthopaedic and Rehabilitation Treatment, Banff, Alberta, Canada, May 25-28, 2016. Paper 0-82, page 69
- [Result] Parent EC, Ghaneei M*, Adeeb S, Schreiber S*, Moreau M, Hedden D, Hill D. (2016). Effects of Schroth exercises added to standard care in adolescents with idiopathic scoliosis (AIS) on marker-less surface topography asymmetry measurements: A randomized controlled trial (RCT) Scoliosis and Spinal Disorders 2017 12(Suppl 1):17 O62. Proceedings of The First Joint Meeting of the International Research Society of Spinal Deformities and the Society on Scoliosis Orthopaedic and Rehabilitation Treatment, Banff, Alberta, Canada, May 25-28, 2016. Paper 0-83, pages 69-70
- [Result] Schreiber S*, Parent E, Khodayari-Moez E, Hedden D, Hill D, Moreau M, Lou E, Watkins E*, Southon S. (2016). Schroth physiotherapeutic scoliosis-specific exercises improve Cobb angles in adolescents with idiopathic scoliosis - A randomized controlled trial. Proceedings of the 10th Annual WCHRI Research Day, Edmonton, Canada, November 16, 2016, Oral 23, page 27
- [Derived] Schreiber S, Parent EC, Hill DL, Hedden DM, Moreau MJ, Southon SC. Patients with adolescent idiopathic scoliosis perceive positive improvements regardless of change in the Cobb angle - Results from a randomized controlled trial comparing a 6-month Schroth intervention added to standard care and standard care alone. SOSORT 2018 Award winner. BMC Musculoskelet Disord. 2019 Jul 8;20(1):319. doi: 10.1186/s12891-019-2695-9. PMID 31286903